CLINICAL TRIAL: NCT04860661
Title: Effect of Prophylactic Esketamine on Postpartum Depression in Cesarean Section: A Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Esketamine on Postpartum Depression in Cesarean Section Women
Acronym: EKET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ailin Luo (Other)
Collaborators: Maternal and Child Health Hospital of Hubei Province (Other); Jingmen No.1 People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Ailin Luo, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EKET
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Esketamine; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The incidence of PPD: the EPDS scale was assessed by face-to-face or telephone interview of the Puerpera 7 d, 30 d, 60 d and 90 d after delivery. EPDS score ≥ 10 was defined as antenatal depression or postpartum emotional disorder.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1. Assign a researcher to determine the order of patients and coordinate the relationship between researchers;
  2. For each patient, an anesthesiologist was assigned to manage anesthesia and collect intraoperative data;
  3. A researcher who was not aware of the protocol was assigned to conduct preoperative evaluation and postoperative follow-up, and received training on evaluation methods before the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N group (Placebo Comparator): 15 minutes after umbilical cord amputation, the patient was intravenously injected with 10 ml normal saline
  Interventions: Drug: Normal saline
- Es group (Experimental): 15 minutes after umbilical cord amputation, the patient was intravenously injected with 0.25mg/kg esketamine, PCIA regimen: sufentanil 100 μ g, esketamine 80 mg, diluted to 100 ml with 0.9% normal saline, set analgesia pump background infusion dose 2 ml/h, single bolus dose 2 ml, locking time 8 minutes.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — After delivery, the parturient was given a loading dose of esketamine, and then a small dose of esketamine was added into PCIA analgesia pump
  Other Names: Es group
  Arms: Es group
Drug: Normal saline — 10 ml normal saline
  Other Names: Ns group
  Arms: N group

SUMMARY:
This study was to explore the preventive effect of esketamine on postpartum depression (PPD) in cesarean section, and to evaluate the safety of the drug

DETAILED DESCRIPTION:
Studies have shown that esketamine can treat clinical refractory depression, the drug takes effect quickly, can quickly eliminate the patient's suicide intention, low-dose maintenance treatment is conducive to the stability of the patient's condition, and less adverse reactions, is the current hot spot of antidepressant drug research. Esketamine has been approved by FDA for the treatment of refractory and suicidal depression, but can it effectively prevent and treat postpartum depression? It is not clear. Based on this, this study aims to explore the preventive effect of prophylactic administration of esketamine on postpartum depression in cesarean section, and evaluate the safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section;
* 18-40 years;
* Primipara;
* Singleton pregnancy;
* Sign informed consent.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) grade III and above;
* Intracranial hypertension;
* Hypertension;
* Severe heart disease;
* Hyperthyroidism patients without treatment or insufficient treatment;
* Liver and kidney dysfunction;
* Preeclampsia or eclampsia;
* Mental disorder, mental retardation;
* Drug abuse and alcoholism;
* Contraindication of intraspinal anesthesia;
* The preoperative EPDS score ≥10;
* Participated in other clinical studies.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The objects of this observation were puerpera with cesarean section
Enrollment: 336 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale(EPDS） scores | up to 90 days after surgery
  EPDS score is 0-30，and ≥ 10 to indicate depression

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) score | 1 Day before operation
  NRS score is 0-10，and ≥ 4 to indicate the pain needs treatment
total number of patient-controlled analgesia (PCA) compressions | up to 24 hours after operation
  the total number of PCA compressions which the patients pressed
total volume of PCA | up to 24 hours after operation
  the total volume of PCA drugs which the patients needed in 24h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ailin luo, Dr., Principal Investigator — Department of Anesthesiology of Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu T, Peng X, Wan K, Li M, Liu T, Shi X, Yao W, Li S, Zhou Z, Yang C, Xu H, Kong J, Wang C, Cheng J, Xu Z, Li D, Liu X, He J, Ye X, Luo A, Xu A, Gao F. Prophylactic esketamine to reduce postpartum depression in primiparae: A multicentre, double-blind, randomised clinical trial. Eur J Anaesthesiol. 2026 Jan 29. doi: 10.1097/EJA.0000000000002348. Online ahead of print. PMID 41607308